CLINICAL TRIAL: NCT06807151
Title: Leveraging Plasma Concentration Levels to Optimize Extracorporeal Treatment in Acute Diquat Poisoning: A Multi-Center Retrospective Cohort Study
Brief Title: Leveraging Plasma Concentration Levels to Optimize Extracorporeal Treatment in Acute Diquat Poisoning
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, Associate Professor, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2023-SR-849
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diquat Poisoning; Blood Purification
Keywords: diquat; poisoning; extracorporeal treatment; hemoperfusion; continuous kidney replacement treatment
MeSH Terms: conditions — Poisoning | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extracorporeal Treatment — Extracorporeal treatments in our study included hemoperfusion and continuous veno-venous hemodiafiltration.

SUMMARY:
This study aimed to evaluate the clinical value of plasma diquat concentration in guiding personalized extracorporeal treatment regimens for patients with acute diquat poisoning.

DETAILED DESCRIPTION:
Diquat (1,1'-ethylene-2,2'-bipyridinium) is a bipyridine herbicide with a structure similar to paraquat. Upon ingestion, diquat induces harmful effects on multiple organ sysmtems, including the gastrointestinal, kidney, liver, musculoskeletal, respiratory, cardiovascular, and central nervous systems. Lethal diquat poisoning primarily manifests as severe toxic encephalopathy and circulatory failure, leading to a high mortality rate. Extracorporeal treatment is widely used in cases of diquat poisoning. ECTRs refer to treatments where toxins are removed outside the body, usually through a circuit. Specifically, ECTRs include hemoperfusion (HP), hemodialysis (HD), continuous kidney replacement treatment (CKRT), extended dialysis, peritoneal dialysis (technically intracorporeal), hemofiltration, hemodiafiltration, therapeutic plasma exchange, and albumin/"liver" dialysis. Several studies have demonstrated that HP can significantly reduce plasma paraquat concentrations, and HP is superior than HD in the clearance of diquat. Additionally, clinical case reports have shown that HP, often combined with CKRT, effectively reduces diquat levels and improves clinical outcomes in patients with diquat poisoning. Continuous veno-venous hemodiafiltration (CVVHDF), a type of CKRT, is primarily used for patients with acute kidney injury (AKI) or fluid overload. The primary goal of CVVHDF is to provide continuous kidney support by removing excess fluids and solutes, there by maintaining electrolyte and acid-base balance. AKI, which is a common consequence of diquat poisoning, impairs kidney function and thus reduces the kidney's ability to clear diquat formula from the plasma. A study reported an AKI incidence of 73.3% in patients with diquat poisoning, indicating many may need CVVHDF. However, the Extracorporeal Treatments in Poisoning (EXTRIP) workgroup does not provide a definitive recommendation on the use of ECTR for diquat poisoning. Aside from case reports and series, there is a lack of evidence to guide clinicians on the optimal application of ECTR in managing diquat poisoning.

ELIGIBILITY:
The inclusion criteria were:

1. history of oral exposure to diquat solution reported by patient or proxy;
2. a specimen for the plasma diquat concentration collected immediately upon admission;
3. documentation that patients or, in case of unconsciousness of the patient, legal proxies were aware of and agreed to treatment plans.

Patients were excluded if:

1. they had ingested other toxins in addition to diquat (qualitative toxicological screening tests);
2. diquat was not detected in specimens, or plasma concentration data were unavailable;
3. patients with an exposure time (time from exposure to presentation) longer than 48 hours;
4. patients had ECTR prior to ED presentation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute diquat poisoning
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
28-day survival | 28 days from the index date
  The primary outcome measure included 28-day survival (survived or died).
Time from exposure to death | 28 days from the index date
  The primary outcome measure included time from exposure to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China